CLINICAL TRIAL: NCT04296240
Title: Safety and Efficacy of Induction and Individualized Neoadjuvant Chemotherapy Based on Oxaliplatin Combined With Fluorouracil for MRF-negative, Moderate-risk and Initially Resectable Middle and Low Rectal Cancer
Brief Title: Induction Chemotherapy for MRF-negative, Moderate-risk, Resectable Middle and Low Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Aiwen Wu, chief, Unit III & Ostomy Service, Gastrointestinal Cancer, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUCH-R03
Record Dates: First submitted 2019-08-26; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; neoadjuvant; chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Antiemetics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemotherapy (Experimental): Oxaliplatin 130mg/m2 d1 and Capecitabine 1250mg/m2 bid1-14 or other fluorouracils, every 21 or 14 days for 2 to 4 cycles, and efficacy evaluation every 2 cycles;
  Interventions: Drug: Oxaliplatin and capecitabine; Procedure: Total Mesorectal Excision

INTERVENTIONS:
Drug: Oxaliplatin and capecitabine — Patients receive 5-Fu and oxaliplatin based neoadjuvant chemotherapy for 3 months
  Other Names: antiemetics
Procedure: Total Mesorectal Excision — Patient receive total mesorectal excision after neoadjuvant chemotherapy
  Other Names: TME

SUMMARY:
This study is designed to test the Safety and efficacy of induction and individualized neoadjuvant chemotherapy based on oxaliplatin combined with fluorouracil for MRF-negative, moderate-risk and initially resectable middle and low rectal cancer.

DETAILED DESCRIPTION:
Preoperative chemoradiation has become standard treatment for stage 2/3 rectal cancer. But for moderate-risk rectal cancer patients, whether neoadjuvant chemotherapy followed with total mesorectal excision is adequate for local control is still unknown. The necessity of preoperative radiotherapy for these patients needs further exploration.

This study is a single-arm, single-center, prospective, phase II clinical study. It is designed to test the efficacy and safety of neoadjuvant chemotherapy for MRF-negative, moderate-risk and initially resectable middle and low rectal cancer.

In this study, patients with MRI defined moderate-risk rectal cancer will receive a three-month neoadjuvant chemotherapy based on Oxaliplatin combined with Fluorouracil(CapeOX,SOX,mFOLFOX6,etc.) and Total mesorectal excision.

Primary Endpoint is pCR rate.Secondary endpoint concludes toxic reactions of neoadjuvant chemotherapy, Incidence of surgical complications and three-year disease-free survival (DFS).

This study is designed to recruit 119 patients in all.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥18 years and ≤80 years

  * ECOG Performance status 0-1
  * Histologically confirmed diagnosis of adenocarcinoma of the rectum
  * The distance from down verge of tumor to anal-rectal junction (ARJ) ≤8cm based on MRI, or ≤12cm based on sigmoidoscopy;
  * Clinical Stage based on MRI

    1. mrMRF(-)
    2. T3c/T3d/T4a, anyN, or T3bN+
  * No evidence of distant metastases
  * No prior pelvic radiation therapy
  * No prior chemotherapy or surgery for rectal cancer
  * No active infections requiring systemic antibiotic treatment
  * ANC > 1.5 cells/mm3, HGB > 10.0 g/dL, PLT > 100,000/mm3, total bilirubin ≤ 1.5 x ULN, AST≤ 3 x ULN, ALT ≤ 3 x ULN.
  * Patients must read, agree to, and sign a statement of Informed Consent prior to participation in this study.

Exclusion Criteria:

* • Recurrent rectal cancer

  * Primary unresectable rectal cancer. A tumor is considered unresectable when invading adjacent organs and an en-bloc resection will not achieve negative margins.
  * The pathological grade was Grade 4, i.e. mucus, signet ring or undifferentiated cancer.
  * Creatinine level greater than 1.5 times the upper limit of normal.
  * Patients who have received prior pelvic radiotherapy.
  * Patients who are unable to undergo an MRI.
  * Patients with a history of a prior malignancy within the past 5 years, except for adequately treated basal cell or squamous cell skin cancer.
  * Patients with a history of any arterial thrombotic event within the past 6 months. This includes angina (stable or unstable), MI, TIA, or CVA.
  * Other Anticancer or Experimental Therapy.
  * Women who are pregnant or breast-feeding.
  * Patients with any other concurrent medical or psychiatric condition or disease which would make them inappropriate candidates for entry into this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response rate | 30 days
  the number of patients with pCR divided by the total number of patients

SECONDARY OUTCOMES:
3 year disease-free survival | three years after the enrollment
  cumulative rate of survival without cancer after 3 years follow up
surgical complication rate | 30 days after the operation
  rate of patients who had surgical complications during the perioperative period
Toxicity of neoadjuvant chemotherapy | 4 months
  category and grade of adverse event during neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Aiwen Wu, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No